CLINICAL TRIAL: NCT03378180
Title: Measurement of Tracheobronchial Tree Using Multiplane CT Reconstructions to Guide Selecting Double-lumen Tubes
Brief Title: Measurement of Tracheobronchial Tree Using 3D CT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Other Study IDs: JHBahk_RUA
Record Dates: First submitted 2017-12-11; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Double Lumen Tube; Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anatomical variations of right main bronchus have been discouraged anesthesiologists' use of right-sided double lumen tubes to facilitate one-lung anesthesia. However, there are absolute indications of right-sided DLTs surgically, such as left pneumonectomy or in cases with left main endobronchial lesions.

With recent advances of 3-dimensional spiral CT reconstruction technique, the investigators conducted this retrospective study to measure accurate length of right and left main bronchus and the angle between the center of the right main bronchus and right upper lobe orifice in axial image to help choosing and further manufacturing right-sided double-lumen tubes.

DETAILED DESCRIPTION:
All CT images will be reviewed using the image measurement software with a slice thickness of 1 mm. A level of -450 Hounsfield units and a width of 1000 Hounsfield units were used for bronchial window settings.

The length of right and left main bronchus will be measured from the tracheal bifurcation to the point of their first branches, respectively, in both 2D- and 3D-CT images. The anteroposterior angulation of right upper lobar bronchus will be measured from the axial 2D-images by the angle between the horizontal midline of the right main bronchus and the center of the RUL orifice which indicates the origin of the RUL bronchus in which the right upper lobar bronchus shows maximal diameter.

ELIGIBILITY:
Inclusion Criteria:

* 3D- thoracic CT scan images obtained between March 1st and October 31th, 2016

Exclusion Criteria:

* younger than 18
* with intraluminal lesions in main bronchus
* with abnormalities of tracheobronchial tree
* with history of tracheobronchial injury or surgery
* diagnosed musculoskeletal deformity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: retrospective measurement of 3D CT scan images obtained from patients admitted for thoracic surgery
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-12-25 (Estimated); Primary Completion 2018-02-20 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
right upper lobe orifice | through study completion, an average of 1 year
  the angle between the center of the right main bronchus and right upper lobe orifice in axial image

SECONDARY OUTCOMES:
length of right and left main bronchus | through study completion, an average of 1 year
  accurate length of both main stem bronchi measured by 3D CT

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea